CLINICAL TRIAL: NCT01393912
Title: Platelet Derived Growth Factor Receptor (PDGFR) Inhibitor Crenolanib in Children and Young Adults With Newly Diagnosed Diffuse Intrinsic Pontine Glioma or Recurrent High-Grade Glioma Including Diffuse Intrinsic Pontine Glioma
Brief Title: PDGFR Inhibitor Crenolanib in Children/Young Adults With Diffuse Intrinsic Pontine Glioma or Recurrent High-Grade Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Arog Pharmaceuticals, Inc. (Industry); The V Foundation for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJPDGF; V Fdn (Other: V Foundation for Cancer Research)
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2016-10

CONDITIONS: Diffuse Intrinsic Pontine Glioma; Progressive or Refractory High-Grade Glioma
Keywords: crenolanib; radiation therapy; malignant brain tumors; pediatric
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Glioma | interventions — crenolanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stratum A Patients (Other): The patients are newly diagnosed Diffuse Intrinsic Pontine Glioma patients. Patients may take crenolanib as an intact tablet or crushed in apple sauce/juice. Currently accruing to dose level 3 (170 mg/m^2).
  Interventions: Drug: Crenolanib
- Stratum B Patients (Other): The patients are recurrent, refractory or progressive high-grade glioma including Diffuse Intrinsic Pontine Glioma patients. Patients may take crenolanib as an intact tablet or crushed in apple sauce/juice. Currently accruing to dose level 4 (220 mg/m^2).
  Interventions: Drug: Crenolanib

INTERVENTIONS:
Drug: Crenolanib — Crenolanib orally administered as whole or crushed tablets once per day with concurrent Radiation Therapy. Crenolanib will continue at the same dose level post Radiation Therapy
  Other Names: CP-868,596

SUMMARY:
This is a Phase I clinical trial evaluating crenolanib (CP-868,596), an inhibitor of Platelet Derived Growth Factor Receptor (PDGFR)-kinase in children and young adults with newly diagnosed diffuse intrinsic pontine glioma (DIPG) (Stratum A) or in recurrent, progressive or refractory High Grade Glioma (HGG) including DIPG (Stratum B). This study drug targets the most commonly amplified region of genome found in DIPG and pediatric high grade glioma (HGG) which encodes for the PDGF receptor kinase. An oral investigational agent crenolanib will be administered daily during and after local radiation therapy (RT) in Diffuse Intrinsic Pontine Glioma DIPG (Stratum A), or daily for children with recurrent/refractory HGG (Stratum B).

DETAILED DESCRIPTION:
Primary Objectives:

* To estimate the maximum tolerated dose (MTD) of crenolanib administered concurrently with RT in pediatric research participants with DIPG
* To estimate the MTD of crenolanib in children and young adults with recurrent/refractory HGG including DIPG
* To characterize the pharmacokinetics of crenolanib in pediatric patients and relate drug disposition to toxicity

Exploratory Secondary Objectives:

* To characterize toxicities and/or adverse events associated with the chronic use of crenolanib
* To evaluate the association between specific polymorphisms of drug metabolizing enzymes and the pharmacokinetics of crenolanib
* To evaluate changes in phosphorylation of targets of PDGF pathway activation in peripheral blood mononuclear cells and investigate the possible relationship between these changes, plasma drug levels of crenolanib and outcome measures
* To evaluate PDGFR, genotype, protein expression and DNA amplification in tumor tissue where available
* To investigate whether magnetic resonance imaging (MRI) techniques that reflect tumor pathophysiology (metabolism, oxygenation, perfusion and vessel wall integrity) are correlated with clinical response
* To characterize the neural tract involvement and tumor progression routes of pediatric brainstem glioma based upon anatomical magnetic resonance imaging and diffusion tensor imaging
* To assess the pattern of failure in radiation therapy in Stratum A participants.
* To describe the research participants' and parents' perspective of symptoms and the quality of life of children enrolled on this phase I trial
* To describe the quality of life and the impact of self-care activities of parents of pediatric research participants enrolled on this phase I trial
* To assess the impact of therapeutic alliance and social support on peace of mind, hope, anxiety/depression and quality of life among parents of pediatric research participants enrolled on this phase I trial

Stratum A- Appropriate dose RT will be administered in 30-33 fractions over approximately 6 weeks for Stratum A patients. Treatment with crenolanib will start on the same day as RT and continue daily during and after Radiation Therapy for a maximum treatment duration of 2 years. We plan to treat a maximum of 5 cohorts of research participants (dosage levels 0, 1, 2, 3, and 4) with escalating doses of crenolanib. A cycle is defined as 28 days and the first 8 weeks of therapy will constitute the dose-limiting toxicity (DLT)-evaluation period.

Stratum B - Crenolanib will be administered orally on a daily basis continuously for 28 days, which defines one cycle. The maximum treatment duration will be 2 years. We plan to treat a maximum of 5 cohorts of research participants (dosage levels 0, 1, 2, 3, and 4) with escalating doses of crenolanib. Dose escalation will be independent of Stratum A escalation. The DLT evaluation period will be four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age must be ≥ 18 months and < or equal to 21 years
* Body surface Area (BSA) ≥ 0.55 m^2
* Lansky (for research participants ≤ 16 years) or Karnofsky (for research participants > 16 years) performance score ≥ 40 at the time of study enrollment
* Adequate organ function at the time of study enrollment as follows:

  * Bone marrow: Absolute neutrophil count (ANC) ≥ 1,000/μL, platelet count ≥ 75,000/μL (transfusion independent), hemoglobin concentration ≥ 8g/dL (may be transfused)
  * Renal: Normal serum creatinine concentration based on age as shown below or glomerular filtration rate (GFR) > 70 ml/min/1.73m^2

    * Age (years): < or equal to 5 and the maximum serum creatinine (mg/dL) is 0.8;
    * 5 < age < or equal to 10 and the maximum serum creatinine (mg/dL) is 1.0;
    * 10< age < or equal to 15 and the maximum serum creatinine (mg/dL) is 1.2;
    * >15 and the maximum serum creatinine (mg/dL) is 1.5;
  * Hepatic: Total bilirubin concentration < or equal to 1.5 times the institutional upper limit of normal for age; SGPT < or equal to 3 times the institutional upper limit of normal
  * Pancreatic: Serum amylase < or equal to 3 times the institutional upper limit of normal for age; lipase < or equal to 3 times the institutional upper limit of normal
* Female research participants of childbearing age must not be pregnant as confirmed by a serum or urine pregnancy test within 1 week of start of treatment. Participants must not be breast-feeding.
* Males or females of reproductive potential may not participate unless they have agreed to use two effective contraceptive methods. Abstinence in a non-sexually active child will be sufficient birth control.

Inclusion Criteria - Stratum A

* Diagnosis of DIPG or high-grade glioma originating from the brainstem.
* Patients have had no previous treatment except corticosteroid use.

Inclusion Criteria - Stratum B

* Patients must have radiologic evidence of recurrent, refractory or progressive high-grade glioma or DIPG. Patients must have either a diagnosis of HGG within the brain and/or spinal cord including DIPG or other high-grade glioma originating from the brainstem. A histologically confirmed diagnosis of anaplastic astrocytoma (WHO grade III), anaplastic oligodendroglioma (WHO grade III), anaplastic oligoastrocytoma (WHO grade III), anaplastic ganglioglioma (WHO grade III), pleomorphic xanthoastrocytoma with anaplastic features (WHO grade III), malignant glioneuronal tumor, glioblastoma multiforme (WHO grade IV) or gliosarcoma (WHO grade IV) is required. For patients with radiologic features of DIPG histologic confirmation of diagnosis is not required.
* Patients must be able to swallow pills or take pills crushed in water based juice or puree (e.g. applesauce, apple juice) by mouth or gastric tube.
* Patients with neurological deficits should have deficits that are stable for a minimum of 1 week prior to registration.
* Patients who are on dexamethasone must be on a stable or decreasing dose for at least one week prior to registration.
* Patients must have fully recovered from the acute toxic effects of chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
* Myelosuppressive chemotherapy: Patients must have received their last dose of known myelosuppressive anticancer chemotherapy at least four weeks prior to study registration or at least six weeks if nitrosourea. At least two weeks must have lapsed if patients received lower dose oral etoposide (50 mg/2) without experiencing evidence of myelosuppression (i.e. neutropenia or requiring transfusion with blood products)
* Biologic agent: Patient must have recovered from any toxicity potentially related to the agent and received their last dose of the biologic agent ≥ 7 days prior to study registration. For biologic agents that have a prolonged half-life, the appropriate interval since last treatment should be discussed with the study chair prior to registration.
* Monoclonal antibody treatment: At least three half-lives must have elapsed prior to registration. Such patients should be discussed with the study chair prior to registration.
* Radiation: Patient has received radiation therapy prior to study registration Patients must have had their last fraction of local irradiation to the primary tumor ≥ 3 months prior to registration and their last fraction of craniospinal irradiation (>24Gy) > or equal to 3 months prior to registration. Patient has not received focal irradiation for symptomatic metastatic sites within 2 weeks prior to registration.
* Bone Marrow Transplant: Patient must be ≥ 3 months since high dose chemotherapy and peripheral blood stem cell rescue prior to registration.
* Growth factors: Patients must be off all colony forming growth factors(s) for at least 1 week prior to registration (filgrastim, sargramostim, erythropoietin) and at least 2 weeks for long-acting formulations (e.g. neupogen).

Exclusion Criteria:

* Metastatic disease outside the CNS.
* Use of enzyme-inducing anticonvulsants (EIACs) within 7 days prior to registration.
* Research participants with uncontrolled infection
* Research participants with any concomitant significant medical illness that in the investigator's opinion cannot be adequately controlled with appropriate therapy, or that would impair the evaluation of side effects related to this treatment, alter drug metabolism or the tolerance to this treatment
* Research participants receiving any other anticancer or investigational drug therapy
* Prior therapy with crenolanib

Of note, the use of any concomitant medication that may affect CYP3A function except for dexamethasone, should be discussed with the principal investigator of this study (or her designee).

Ages: 18 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2011-07; Primary Completion 2014-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Estimate the maximum tolerated dose (MTD) of crenolanib in pediatric research participants with newly diagnosed DIPG | 2.5 years
  This is done using rolling 6 -design
Estimate the MTD of crenolanib in children and young adults with recurrent/refractory HGG including DIPG | 2.5years
  This is done using rolling 6 design
Characterize the pharmacokinetics of crenolanib in pediatric patients and relate drug disposition to toxicity | 2.5 years
  Individual pharmacokinetic parameters will be estimated using nonlinear mixed effects modeling methods (NONMEM) to estimate both the inter- and intra-subject variability.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Broniscer, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols